CLINICAL TRIAL: NCT07008859
Title: Correlation Between Voice Pitch Changes and Tension of Suboccipital Muscles In Normal Subjects
Status: Active, not recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Basant Sabry Mohamed Elbana, physiotherapist, Cairo University
Other Study IDs: 012/005045
Record Dates: First submitted 2025-05-21; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-04

CONDITIONS: Voice Change; Suboccipital Muscles Tension
Keywords: voice pitch changes; tension of suboccipital muscles; correlational study
MeSH Terms: conditions — Dysphonia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
this study for investigation of correlation between voice pitch and tension of suboccipital muscles

DETAILED DESCRIPTION:
participants will be assigned randomly , normal people i will use 2 instruments first : compturized speech lab (CSL) to analyze voice pitch second: electromyography EMG to measure suboccipital muscle tension during speech this task will be repated twice first one during normal speech , second one during change in voice pitch

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 20-60 years.
* No history of musculoskeletal disorders, voice disorders, or neurological conditions.
* Normal voice function (Voice Handicap Index [VHI]-10 ≤ 11) .

Exclusion Criteria:

* Individuals with neck pain or injury in the past six months.
* History of vocal pathologies, recent surgeries, or auditory impairments

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: participatnts are normal people ,both gender , aged 20-60 years . number of participants are 119
Sampling Method: Probability Sample
Enrollment: 119 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
tension of suboccipital muscles | immediately during voice pitch changes

SECONDARY OUTCOMES:
suboccipital muscles tension | 5 minutes :tension will be measured twice during speech
  suboccipital muscles tension will be measured by Electromyography during change of voice pitch

CONTACTS AND LOCATIONS:
Overall Officials: basant sabry elbana, bachelor of physical therapy, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy , Cairo University, Dokki, Egypt, Egypt